CLINICAL TRIAL: NCT06714994
Title: Effect of Spectacle Distribution to Myopic Secondary School Students in Rural Communities of Liaoning Province on Communities Academic High School Enrolment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SWISH
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Children at Intervention schools will receive free spectacles of a design they select, based on the child's measured refractive power and dispensed at school by the teacher. All students will be advised to wear glasses as much as possible during the study to ensure clear vision.
  Interventions: Device: free spectacles
- Control group (No Intervention): Children at Control schools will receive a glasses prescription and letter to the parents informing them of the refractive status of their child, with free glasses provided only at the end of the trial. Service offered to the Control group exceeds standard care, in that no school-based programs of vision screening and refraction currently exist in the study area, or in most of rural China.

INTERVENTIONS:
Device: free spectacles — Children will receive free spectacles
  Arms: Study group

SUMMARY:
To determine whether provision of free spectacles to rural-dwelling Chinese secondary school students with visually-significant refractive error, together with a teacher-based incentive to promote their use, increases the proportion of children going on to academic high school, as opposed to dropping out or pursuing a vocational track.

DETAILED DESCRIPTION:
The investigators propose in the current trial to significantly expand the evidence base for spectacle distribution as the most-effective health intervention to improve educational opportunities for China's under-served rural children and adolescents by assessing impact on school attainment.

ELIGIBILITY:
Inclusion Criteria:

* Year 1 students (about 12-15 years old) from schools in county-level cities and below in Liaoning Province
* Uncorrected (self-glasses) visual acuity of ≤6/12 in both eyes
* Refractive error meets cut-offs shown to be associated with significantly greater improvement in visual acuity when corrected7 (myopia ≤-0.75 diopters (D, or astigmatism (non-spherical refractive error) ≥1.00 D
* Best corrected visual acuity ≥6/7.5 in either eye

Exclusion Criteria:

* Hyperopia ≥2.00 D
* Presence of visually-significant ocular condition besides refractive error

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1980 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Attendance at academic high school | In July following completion of Year 3 of Middle School. This occurs after 32 months of participant followup.
  This will be assessed by systematically contacting parents, teachers and students to ascertain enrolment status, which REAP has used to obtain > 97% follow-up in previous studies of high school accession. In the event of inconsistent responses, priority will be given to responses of parents, then teachers and finally students

SECONDARY OUTCOMES:
Compliance with spectacle wear | After 12 months of participant followup
  Actual presence of spectacles on the child's face (rather than having glasses at school)at the time of an unannounced examination.
Classroom use of blackboards versus textbooks | After 12 months of participant followup
  Frequency of blackboard versus textbook use in the major subjects (Maths Chinese, English) on a questionnaire administered to teachers, and answered as "all", "most", "about half", little" or "none" of teaching.
Cost effectiveness of intervention. | At study closeout, after 32 months of participant follow up
  Calculated as ratio of incremental cost to proportion of children who continue to academic high school as opposed to vocational high school or no schooling. Incremental cost is the difference of costs between implementation of intervention and control, Intervention costs will comprise the screening test glasses (including replacements).
Depression and Anxiety | At baseline and 12 months post-treatment
  Depression and anxiety score measured with Anxiety Stress Scale (DASS). The score range for depression, anxiety and stress are 0-42, with higher score indicates more severe mental health problems.
Self Esteem | At baseline and 12 months post-treatment
  Self-esteem score measured with the Rosenberg Self-esteem Scale. The scores range from 0-30, with higher scores indicate higher self-esteem.
Emotional and behavioral problems | At baseline and 12 months post-treatment
  Emotional and behavioral problems score using the Strengths and Difficulties Questionnaire (SDQ), with difficulties score ranges from 0 to 40, Prosocial scale ranges from 0-10,with higher score indicates severe mental health and behavioral problems.
Progression of Shortsightedness | At baseline and 12 months post-treatment
  Progression of Shortsightedness will be measured using change in refraction over time

CONTACTS AND LOCATIONS:
Overall Officials: Guanghao Qin, Study Chair — He Eye Hospital
Locations (1):
- He Eye Specialist Hospital, Shenyang, China

IPD SHARING:
Plan to Share IPD: No
Anonymized datasets generated and analyzed during the current study will be made available on reasonable request by the PI

REFERENCES:
- [Background] Ma X, Zhou Z, Yi H, Pang X, Shi Y, Chen Q, Meltzer ME, le Cessie S, He M, Rozelle S, Liu Y, Congdon N. Effect of providing free glasses on children's educational outcomes in China: cluster randomized controlled trial. BMJ. 2014 Sep 23;349:g5740. doi: 10.1136/bmj.g5740. PMID 25249453
- [Background] Ma Y, Congdon N, Shi Y, Hogg R, Medina A, Boswell M, Rozelle S, Iyer M. Effect of a Local Vision Care Center on Eyeglasses Use and School Performance in Rural China: A Cluster Randomized Clinical Trial. JAMA Ophthalmol. 2018 Jul 1;136(7):731-737. doi: 10.1001/jamaophthalmol.2018.1329. PMID 29801081
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Jiang C, Zhu Y, Luo Y, Tan CS, Mastrotheodoros S, Costa P, Chen L, Guo L, Ma H, Meng R. Validation of the Chinese version of the Rosenberg Self-Esteem Scale: evidence from a three-wave longitudinal study. BMC Psychol. 2023 Oct 18;11(1):345. doi: 10.1186/s40359-023-01293-1. PMID 37853499
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702